CLINICAL TRIAL: NCT05152537
Title: A Multicenter Prospective Cohort Study of FLOR3 Gene Polymorphism in Predicting Outcomes of TKI-stopping in Chronic Myeloid Leukemia
Brief Title: FLOR3 Gene Polymorphism in Predicting Outcomes of Tyrosine Kinase Inhibitor（TKI）Stopping in Chronic Myeloid Leukemia
Acronym: NTU-CML-001
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: AHNTU-CML-001
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-08

CONDITIONS: Folate; CML; Treatment-free Remission
Keywords: FOLR3; CML; TFR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5ml Peripheral blood of CML patients who discontinued TKI treatment are extracted and stored.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For patients with chronic myeloid leukemia in chronic phase (CML-CP) who have achieved a stable deep molecular response (DMR) using BCR-ABL1 tyrosine kinase inhibitors (TKIs), treatment-free remission (TFR) following TKI cessation is an emerging goal. However, about half of the patients relapsed after TKI discontinuation. There is no definite examinations to predict the outcome of TKI discontinuation. Investigators aim to study the relationship between FLOR3 SNP rs139130389 and the outcome of TKI discontinuation.

DETAILED DESCRIPTION:
Investigators aim to detect FOLR3 SNP rs139130389, and establish its correlation with patients' treatment response, remission time, TKI resistance and the outcome of TKI stopping.

ELIGIBILITY:
Inclusion Criteria:

1. The patient signs the informed consent form
2. Age over 18, male or female
3. The patient was diagnosed as chronic phase of CML.
4. ECoG score 0-2
5. Receive TKI treatment for at least 4 years and continuously obtain MR4 or mr4.5 for at least 3 years.
6. The subjects fully understand and comply with the requirements of the research scheme and are willing to complete the research as planned.

Exclusion Criteria:

NA

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. The patient signs the informed consent form
  2. Age over 18, male or female
  3. The patient was diagnosed as chronic phase of CML.
  4. ECoG score 0-2
  5. Receive TKI treatment for at least 4 years and continuously obtain MR4 or mr4.5 for at least 3 years.
  6. The subjects fully understand and comply with the requirements of the research scheme and are willing to complete the research as planned.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
treatment-free remission or relapse | 1 year
  Observe whether the patients were in remission or relapse 1 year after drug withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, Doctorate, Study Chair — Affiliated Hospital of Nantong University
Locations (1):
- Affliated Hospital of Nantong University, Nantong, China

IPD SHARING:
Plan to Share IPD: No